CLINICAL TRIAL: NCT01588600
Title: Effects of Fiber on Satiety and Food Intake in Men and Women
Brief Title: Effects of Fiber on Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ingredion Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: UL001
Record Dates: First submitted 2012-04-10; First posted 2012-05-01 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2012-04

CONDITIONS: Obesity
Keywords: food intake, satiety, fiber
MeSH Terms: conditions — Obesity | interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Breakfast without fiber
  Interventions: Other: Dietary Fiber
- Low-dose (Experimental): Low-dose of fiber in breakfast
  Interventions: Other: Dietary Fiber
- High-dose (Experimental): high dose of fiber added to breakfast
  Interventions: Other: Dietary Fiber

INTERVENTIONS:
Other: Dietary Fiber — Fiber added to breakfast

SUMMARY:
The effects of a dietary fiber on hunger and food intake will be tested in men and women. Participants will receive fiber as part of a breakfast meal on two occasions. On another occasion, participants will receive the same breakfast, without added fiber. Their feelings of hunger and fullness will be measured over the day. They will be offered lunch, dinner and an evening snack and how much they eat will be recorded. It is expected that the fiber supplement will enhance their feelings of satiety and reduce the amount they eat over the day.

ELIGIBILITY:
Inclusion Criteria:

* normal-weight adults

Exclusion Criteria:

* eating disorders,
* on medications that affect food intake,
* pregnant or lactating,
* non-breakfast eaters

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Food intake | 24-hr food intake, on three occasions within 3 weeks
  24-hour Food intake will be measured 3 times

SECONDARY OUTCOMES:
Subjective appetite ratings | Hourly, over 8 hrs, on 3 days within a 3-week period
  Ratings of hunger and fullness will be assessed 18 times

CONTACTS AND LOCATIONS:
Overall Officials: Jason Halford, PhD, Principal Investigator — University of Liverpool
Locations (1):
- Kissileff Laboratory for the Study of Human Ingestive Behavior, Liverpool, United Kingdom